CLINICAL TRIAL: NCT06183034
Title: The Study of Acceptability and Feasibility of a Preoperative Very Low Calorie Diet Intervention on Surgical Weight Loss Outcomes (SAFETY)
Brief Title: Acceptability and Feasibility of a Preoperative Very Low Calorie Diet Intervention on Surgical Weight Loss Outcomes (SAFETY)
Acronym: SAFETY
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Hartford Hospital (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: R-HHC-2023-0179
Record Dates: First submitted 2023-12-13; First posted 2023-12-27 (Actual); Last update posted 2024-02-28 (Actual); Status verified 2023-11

CONDITIONS: Obesity
MeSH Terms: conditions — Obesity

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Very Low Calorie Diet (Other): Very Low Calorie Diet - caloric intake restricted to approximately 800 kcal/day
  Interventions: Other: Very Low Calorie Diet

INTERVENTIONS:
Other: Very Low Calorie Diet — Participants will receive a very low calorie diet as described in the arm/group

SUMMARY:
Class 4 obesity is defined as a BMI ≥50Kg/m2, representing approximately ≥150 pounds of excess weight. For patients with Class 4 obesity, metabolic and bariatric surgery (MBS) is the only effective treatment. However, MBS is associated with a higher rate of perioperative morbidity and mortality for patients with Class 4 obesity. Additionally, more patients with Class 4 obesity experience suboptimal weight loss. For patients with Class 4 obesity, preoperative weight loss can reduce the technical difficulty of surgical procedures, rendering MBS safer. Preoperative weight loss may also decrease visceral adipose tissue and liver volume as well as reduce weight-related comorbidities.

A very low-calorie diet (VLCD), which involves restricting caloric intake to approximately 800 kcal/day, is one strategy to help patients achieve weight loss preoperatively. Although studies show that a VLCD prior to MBS yields weight loss, reduces liver volume and rates of perioperative complications, most preoperative VLCDs are short (2-8 weeks) with variable adherence. To date, no study has systematically assessed the feasibility and acceptability of a standard 12-week VLCD among patients with BMI ≥50 pursuing MBS. No study has evaluated postoperative weight loss among patients who have undergone a preoperative VLCD.

This study will be a single arm trial designed to test the feasibility, acceptability, and preliminary efficacy of a 12-week VLCD program prior to sleeve gastrectomy (SG) and associated weight loss up to 1 year following MBS. The investigators will enroll 24 patients aged 18-70, with a BMI≥50Kg/m2, and are approved for SG. Participants will consume up to 5 meal replacement protein shakes and 2 cups of vegetables daily for 12 weeks. Participants will attend weekly in-person office visits with the clinicians at the Hartford Hospital Medical and Surgical Weight Loss Center in Glastonbury, CT to assess weight loss, physical and mental health, feasibility and acceptability of and adherence to the VLCD. The investigators hypothesize that a 12-week VLCD is feasible in this population, defined as ≥70% (18 out of 24 participants) completing the program. The investigators hypothesize that better attendance at the weekly visits and higher adherence to the diet recommendations will provide greater weight loss preoperatively and percent total weight loss at the completion of VLCD, on the day of MBS, and at 3, 6, and 12 months post-surgery. Findings from this study may lead to additional projects that aim to develop and implement an optimal pre-surgery and post-surgery clinical care model for bariatric patients.

ELIGIBILITY:
Inclusion Criteria:

* BMI greater than or equal to 50 kg/m2
* Eligible and approved for sleeve gastrectomy as primary bariatric treatment (eligibility and approval for sleeve gastrectomy will be determined from a surgical standpoint by the surgeon)
* Able and willing to sign an Informed Consent document

Exclusion Criteria:

* Qualified for Roux-en-Y gastric bypass
* On FDA-approved weight loss medications at time of consult
* Are lactose intolerant
* History of Type 1 diabetes
* Have had lap band or other prior bariatric surgery
* Global functioning score (GFR) ≤45 mL/min/1.73 m² (this is assessed as a part of the routine procedure for all patients)
* >70 years old (our program does surgery on very few patients over this age)
* Weight is above 300 kgs (~660 lbs.). (The weight limit for SECA scales is 300 kgs maximum).
* Have been diagnosed with end stage renal disease (CKD stage 3-5) and on dialysis
* Severe depression measured by Beck Depression Inventory (BDI) (BDI score greater than or equal to 30)
* History of severe psychiatric disorder (schizophrenia, schizoaffective, or bipolar disorder)

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Estimated)
Dates: Start 2024-03-05 (Estimated); Primary Completion 2025-10-31 (Estimated); Study Completion 2025-12-30 (Estimated)

PRIMARY OUTCOMES:
Percentage of participants who complete the 12-week VLCD program | Week 1 through 12 of the 12 week VLCD program
  Completion is defined as attendance at 10 or more weekly visits, including the week 12 visit

SECONDARY OUTCOMES:
Consumption of 3-5 meal replacement shakes plus 2 cups of vegetables per day for 5 to 7 days | Measured every day of 12 week VLCD program
VLCD acceptability | data collected at week 1, week 6, and week 12 of VLCD program
  Acceptability will be measured using a sum of 8 items on a survey with eight 5-point Likert scale questions (e.g., I find the VLCD meal plan easy to follow) on a scale from 1 [strongly disagree] to 5 [strongly agree]). VLCD acceptability is defined as ≥75% of the participants having a mean survey rating of ≥4.

OTHER OUTCOMES:
Weight in pounds | Measured on the day of bariatric surgery and at 3, 6, and 12 month post-surgery follow up visit

CONTACTS AND LOCATIONS:
Locations (1):
- Hartford Hospital, Hartford, Connecticut, United States

IPD SHARING:
Plan to Share IPD: No